CLINICAL TRIAL: NCT03522844
Title: Comparative Effectiveness of Mindfulness-Based Stress Reduction and Pharmacotherapy for Anxiety
Brief Title: Treatments for Anxiety: Meditation and Escitalopram
Acronym: TAME
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Elizabeth Hoge, Principal Investigator, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-1464
Record Dates: First submitted 2018-05-01; First posted 2018-05-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Anxiety Disorders; Generalized Anxiety Disorder; Panic Disorder; Social Anxiety Disorder; Agoraphobia
Keywords: mindfulness; escitalopram; anxiety
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder; Panic Disorder; Phobia, Social; Agoraphobia | interventions — Mindfulness-Based Stress Reduction; Escitalopram

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive one of two treatments over the course of 8-weeks. One group will participate in an 8-week Mindfulness-Based Stress Reduction Course and the other group will receive a daily medication treatment (escitalopram).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Mindfulness-Based Stress Reduction (MBSR) (Experimental)
  Interventions: Other: Mindfulness-Based Stress Reduction
- Escitalopram (Active Comparator)
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Other: Mindfulness-Based Stress Reduction — Participants randomized to the MBSR intervention will consist of an 8-week Mindfulness-Based Stress Reduction (MBSR) program, taught and facilitated by a trained instructor. The classes instruct participants in the theory and practice of several forms of mindfulness meditation: a body scan, breathing awareness, and mindfulness stretching exercises designed to bring awareness of the body and current experience of movement. The intervention will include a weekly class for 8 weeks and classes will be 2.5 hours in duration. The intervention will also include a 1-day (7 hours) retreat on a weekend at the end of the program. Participants will also be asked to engage in 45 minutes of practice at home on a daily basis, as well as informal practice assignments that instruct participants to bring mindfulness to current daily activities.
  Arms: Mindfulness-Based Stress Reduction (MBSR)
Drug: Escitalopram — Escitalopram is an antidepressant, widely used to treat anxiety disorders. During the 8 weeks of randomized treatment with escitalopram, subjects will be seen regularly by a study physician. The pill medication will be initiated at 10 mg/day; at week 2, dosage will be increased to 20 mg/day if well tolerated (or delayed if not). Side effects will be assessed at each visit and recorded.
  Arms: Escitalopram

SUMMARY:
We propose the first randomized, controlled study to assess the comparative effectiveness of Mindfulness-Based Stress Reduction (MBSR) with a medication for anxiety disorders. We will use escitalopram, gold-standard SSRI treatment for patients with anxiety disorders, and will examine the comparative effectiveness of the two treatments on anxiety symptoms and other outcomes important to patients.

DETAILED DESCRIPTION:
Mindfulness meditation treatments have been growing in popularity and becoming widely disseminated, and people with anxiety are interested in mindfulness. A benefit of mindfulness interventions is that they can be provided outside of a mental health setting, which may make them more acceptable to patients. Although mindfulness meditation is gaining popularity, there is no information how this treatment strategy compares with standard treatment, such as with medication. Patients need more information about the comparison of treatments to be able to make informed decisions about their health care. We propose the first randomized, controlled study to assess the comparative effectiveness of Mindfulness-Based Stress Reduction (MBSR) compared to escitalopram, a standard medication for patients with anxiety disorders such as generalized anxiety disorder, social anxiety disorder, panic disorder, and agoraphobia.

Patients will be randomized into two 8-week treatments: (1) MBSR and (2) escitalopram. To enroll the necessary sample, we will utilize three study sites in different geographic locations that each have strong clinical and research infrastructures: Georgetown University Medical Center, Massachusetts General Hospital and New York University Langone Medical Center. Thus, we will take advantage of three productive teams with previous successful collaborations and experience in mind-body treatment studies.

Adaptations and Additional Aims:

Due to the COVID-19 pandemic, the study was transitioned to a virtual format (on-line videoconference visits) in March 2020 as a pilot adaptation with the introduction of additional aims to explore the following: (1) the comparative effectiveness and treatment satisfaction for in-person MBSR versus virtual MBSR and (2) the comparative effectiveness of virtual MBSR versus virtual pharmacotherapy. An additional 202 participants were randomized to the virtual version of the study to support these aims.

Note about the in-person recruitment: Due to the impact of pandemic-related and participant-related confounders, it has not been possible to return to in-person treatments since March 2020. Before the pandemic, we had published a methods paper adopting (a priori) a non-inferiority margin of 0.495 points on the CGI-S for the analysis of the primary hypothesis. Although we were not able to enroll the proposed sample size of 368 due to the pandemic, with 276 patients randomized, we have sufficient statistical power of 80% for our original analysis to stop in person enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between 18 and 75 years old.
2. Have an anxiety disorder, including: social anxiety disorder (SAD), generalized anxiety disorder (GAD), panic disorder, or agoraphobia
3. Must understand study procedure and be willing to participate in all testing visits and treatment as assigned.
4. Participants must be able to give informed consent to the study procedures.

Exclusion Criteria:

1. Comorbid psychiatric disorder other than anxiety or depression, such as psychotic disorder, post-traumatic stress disorder, obsessive compulsive disorder, eating disorders, bipolar disorder; developmental or organic mental disorders; and current (past 6 months) substance use disorders.
2. A serious medical condition that may result in surgery or hospitalization.
3. A history of head trauma causing loss of consciousness, or ongoing cognitive impairment
4. Inability to understand study procedures or informed consent process, or significant personality dysfunction likely to interfere with study participation (assessed during the clinical interview).
5. Subjects who will be non-compliant with the study procedures. This may include planned travel out of town.
6. Pregnancy as assessed by urine test at screen. Avoidance of pregnancy is also necessary for inclusion in the study.
7. Subjects taking barbiturates, SSRIs, anti-depressants, or antipsychotics. Sleep medications (other than anti-depressants) and benzodiazepines will be allowed, if has been taken at stable dose 4 weeks prior to baseline and the patient plans to continue at the same dose through the trial. Trazadone (for sleep) above 100mg will be disallowed.
8. Concurrent psychotherapy initiated within 1 month of screen interview, or ongoing psychotherapy of any duration directed specifically toward the treatment of anxiety (such as cognitive behavioral therapy).
9. Individuals who have completed a course of MBSR or an equivalent meditation training in the last year, or have an ongoing daily meditation practice
10. Individuals reporting significant active suicidal ideation or suicidal behaviors within the past year.
11. Individuals with a medical condition (i.e., epilepsy) that may be exacerbated by study treatment, as determined by a study physician or nurse practitioner based on history, physical, and/or labs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression of Severity scale | 8 weeks
  The CGI is a measure of symptom severity and is rated by a clinician

SECONDARY OUTCOMES:
Clinical Global Impression- Improvement (CGI-I) | 8 weeks
  The CGI-I measures symptom improvement and is rated by a clinician
Structured Interview Guide for the Hamilton Anxiety Scale (SIGH-A) | 8 weeks
  The SIGH-A assesses general anxiety symptoms and is rated by a clinician
Liebowitz Social Anxiety Scale (LSAS) | 8 weeks
  The LSAS measures social anxiety and is rated by a clinician
Panic Disorder Severity Scale (PDSS) | 8 weeks
  The PDSS measures panic symptom severity and is rated by a clinician
Overall Anxiety Severity and Impairment Scale (OASIS) | 8 weeks
  The OASIS is a patient-reported measure is anxiety symptoms
Pittsburgh Sleep Quality Index (PSQI) | 8 weeks
  The PSQI is a patient-reported measure of sleep
Penn State Worry Questionnaire (PSWQ) | 8 weeks
  The PSWQ is a patient-reported measure of worry
Beck Anxiety Inventory (BAI) | 8 weeks
  The BAI is a patient-reported measure is anxiety symptoms
PROMIS-Satisfaction with Participation in Social Roles (SPSR) | 8 weeks
  The PROMIS-SPSR is a patient-reported measure of contentment with social roles
PROMIS- Emotional Distress Scales (ED) | 8 weeks
  The PROMIS-ED scales are patient-reported measures of emotional distress, such as anxiety and depression
PROMIS-Ability to Participate in Social Roles and Activities (APSRA) | 8 weeks
  The PROMIS-APSRA is a patient-reported measure of ability to perform usual social roles and activities

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Massachusetts General Hospital, Boston, Massachusetts
  - New York University, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hoge EA, Mete M, Baker AW, Szuhany KL, Armstrong CH, Steinberg MH, Dutton MA, Bui E, Simon NM. A randomized controlled trial comparing mindfulness to escitalopram for anxiety: In-person and remote, synchronous delivery pre and post COVID-19 pandemic. J Affect Disord. 2025 Sep 1;384:163-172. doi: 10.1016/j.jad.2025.04.145. Epub 2025 May 3. PMID 40324655
- [Derived] Hu H, Mete M, Rustgi NK, Washington CI, Sanghavi K, Dutton MA, Simon NM, Baker AW, Bui E, Hoge EA. Mindfulness Meditation vs Escitalopram for Treatment of Anxiety Disorders: Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2024 Oct 1;7(10):e2438453. doi: 10.1001/jamanetworkopen.2024.38453. PMID 39382900
- [Derived] Oft AC, Philip S, Holz E, Sathi S, Geng X, Hoge E. Effect of meditation or escitalopram on work performance in patients with anxiety disorders. J Affect Disord. 2024 Nov 1;364:104-107. doi: 10.1016/j.jad.2024.08.019. Epub 2024 Aug 10. PMID 39134156
- [Derived] Hoge EA, Bui E, Mete M, Dutton MA, Baker AW, Simon NM. Mindfulness-Based Stress Reduction vs Escitalopram for the Treatment of Adults With Anxiety Disorders: A Randomized Clinical Trial. JAMA Psychiatry. 2023 Jan 1;80(1):13-21. doi: 10.1001/jamapsychiatry.2022.3679. PMID 36350591